CLINICAL TRIAL: NCT03474484
Title: Calprotectin I in Serum as a Diagnostic Marker of Pneumonia in Patients Hospitalised With Acute COPD Exacerbation
Brief Title: Calprotectin I Serum as a Diagnostic Marker
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 20171496/REK midt
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Biomarkers; Sensitivity and Specificity; Clinical Deterioration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypersensitivity; Clinical Deterioration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The standard hospital procedures were followed for collection and processing of blood for the analysis of C-reactive protein (CRP) and white blood cell count (WBC). Additional blood samples for calprotectin were obtained at admission (T0) and 6 (T1), 24 (T2) and 48 (T3) hours post admission. Serum specimens for the calprotectin analysis were stored at minus 70°C until they were analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- np-AECOPD: Patients with evidence of acute exacerbation of chronic obstructive pulmonary disorder (AECOPD) and pulmonary infiltrate on chest X -ray at admission
- p-AECOPD: Patients with evidence of acute exacerbation of chronic obstructive pulmonary disorder (AECOPD) without pulmonary infiltrate on chest X -ray at admission

SUMMARY:
Lower respiratory tract infection is the most common cause of acute exacerbations of chronic obstructive pulmonary disease (AECOPD). Patients diagnosed with pneumonia in addition to an AECOPD experience more severe clinical and laboratory disease manifestations, increase in-hospital morbidity and worse outcome. Clinicians have sought for new biomarkers that together with clinical assessments can improve the diagnostic accuracy of pneumonia in patients with AECOPD.The aim of the present study is to compare the accuracy of calprotectin with procalcitonin (PCT), C-reactive protein (CRP) and white blood cell count (WBC).

ELIGIBILITY:
Inclusion Criteria:

* clinically confirmed acute exacerbation of chronic obstructive pulmonary disorder (AECOPD)
* COPD diagnosis previously confirmed by spirometry according to the GOLD criteria.

Exclusion Criteria:

* known malignant disease
* bronchiectasis
* chronic bacterial colonisation of the airways
* treatment with an immunosuppressive drug or long-term treatment with antibiotics.
* not examined with a chest X-ray at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Thoracic Medicine at Trondheim University Hospital (TUH) due to an AECOPD, age > 18years old. (EU). The patients were examined at the Emergency Unit and included in the study if they had a COPD diagnosis previously confirmed by spirometry according to the GOLD criteria and a clinically confirmed AECOPD
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Calprotectin concentration in serum | Change in serum concentration from baseline to 48 hours
  ELISA-kit (MRP8/14 ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Anne h. Henriksen, md phd, Study Director — St Olavs Hospital HF
Locations (1):
- Department of Thoracic and Occupational Medicine, Trondheim, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the requirements from journal where results of this study will be published

REFERENCES:
- [Background] Titova E, Aune MW, Fonn K, Henriksen AH, Asberg A. Neutrophil CD64 Expression as a Diagnostic Marker in Patients Hospitalized with Exacerbations of COPD: A Prospective Observational Study. Lung. 2015 Oct;193(5):717-24. doi: 10.1007/s00408-015-9762-2. Epub 2015 Jul 15. PMID 26174093